CLINICAL TRIAL: NCT05257083
Title: A Phase 3 Randomized Study Comparing Daratumumab, Bortezomib, Lenalidomide and Dexamethasone (DVRd) Followed by Ciltacabtagene Autoleucel Versus Daratumumab, Bortezomib, Lenalidomide and Dexamethasone (DVRd) Followed by Autologous Stem Cell Transplant (ASCT) in Participants With Newly Diagnosed Multiple Myeloma Who Are Transplant Eligible
Brief Title: A Study of Daratumumab, Bortezomib, Lenalidomide and Dexamethasone (DVRd) Followed by Ciltacabtagene Autoleucel Versus Daratumumab, Bortezomib, Lenalidomide and Dexamethasone (DVRd) Followed by Autologous Stem Cell Transplant (ASCT) in Participants With Newly Diagnosed Multiple Myeloma
Acronym: CARTITUDE-6
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Stichting European Myeloma Network (Network)
Collaborators: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Organization: European Myeloma Network B.V. (Network)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EMN28/68284528MMY3005; 2021-003284-10 (EudraCT Number)
Record Dates: First submitted 2022-02-16; First posted 2022-02-25 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Multiple Myeloma
Keywords: Cellular Therapy; CAR-T Therapy; BCMA CAR-T; Newly Diagnosed Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — daratumumab; Bortezomib; Lenalidomide; Dexamethasone; Cyclophosphamide; fludarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Arm A: DVRd + ASCT+DVRd (Standard Therapy) (Active Comparator): Participants will receive daratumumab, bortezomib, lenalidomide and dexamethasone (DVRd) for 4 induction cycles. Followed by ASCT and 2 cycles of DVRd consolidation, and lenalidomide maintenance therapy for 2 years
  Daratumumab subcutaneously (SC), 1800 mg on days 1, 8, 15 and 22 of cycle 1 and 2, on days 1 and 15 of cycle 3-6.
  Bortezomib SC 1.3 mg/m^2 on days 1, 4, 8, and 11 of each cycle 1-6. Lenalidomide orally, 25 mg on days 1 to 21 of each cycle 1-6. Dexamethasone orally, 40 mg once a week on days 1, 8, 15 and 22 of each cycle 1-6.
  Each cycle will consist 28 days.
  Lenalidomide maintenance orally 10 to 15 mg on days 1 to 28 (continuously) until confirmed progressive disease or unacceptable toxicity or for a maximum of 2 years
- Arm B: DVRd followed by Ciltacabtagene Autoleucel (Experimental): Participants will receive daratumumab, bortezomib, lenalidomide and dexamethasone (DVRd) for 6 induction cycles.
  Participants will receive a conditioning regimen (cyclophosphamide 300 mg/m^2 intravenous [IV] and fludarabine 30 mg/m^2 IV daily for 3 days) and Cilta-cel infusion 0.75*10^6 chimeric antigen receptor (CAR)-positive viable T cells/kilogram (kg), followed by lenalidomide post CAR-T cell therapy for 2 years
  Daratumumab subcutaneously (SC), 1800 mg on days 1, 8, 15 and 22 of cycle 1 and 2, on days 1 and 15 of cycle 3-6.
  Bortezomib SC 1.3 mg/m^2 on days 1, 4, 8, and 11 of each cycle 1-6.
  Lenalidomide orally, 25 mg on days 1 to 21 of each cycle 1-6.
  Dexamethasone orally, 40 mg once a week on days 1, 8, 15 and 22 of each cycle 1-6.
  Each cycle will consist of 28 days.
  Lenalidomide maintenance orally 10 to 15 mg on days 1 to 28 (continuously) until confirmed progressive disease or unacceptable toxicity or for a maximum of 2 years
  Interventions: Drug: Daratumumab; Drug: Bortezomib; Drug: Lenalidomide; Drug: Dexamethasone; Drug: Cilta-cel; Drug: Cyclophosphamide; Drug: Fludarabine

INTERVENTIONS:
Drug: Daratumumab — Daratumumab will be administered SC.
  Arms: Arm B: DVRd followed by Ciltacabtagene Autoleucel
Drug: Bortezomib — Bortezomib will be administered SC.
  Arms: Arm B: DVRd followed by Ciltacabtagene Autoleucel
Drug: Lenalidomide — Lenalidomide will be administered orally.
  Arms: Arm B: DVRd followed by Ciltacabtagene Autoleucel
Drug: Dexamethasone — Dexamethasone will be administered orally.
  Arms: Arm B: DVRd followed by Ciltacabtagene Autoleucel
Drug: Cilta-cel — Cilta-cel will be administered intravenously
  Other Names: JNJ-68284528
  Arms: Arm B: DVRd followed by Ciltacabtagene Autoleucel
Drug: Cyclophosphamide — Cyclophosphamide will be administered intravenously.
  Arms: Arm B: DVRd followed by Ciltacabtagene Autoleucel
Drug: Fludarabine — Fludarabine will be administered intravenously.
  Arms: Arm B: DVRd followed by Ciltacabtagene Autoleucel

SUMMARY:
The purpose of this study is to compare the efficacy of Daratumumab, Bortezomib, Lenalidomide and Dexamethasone (DVRd) followed by Ciltacabtagene Autoleucel versus Daratumumab, Bortezomib, Lenalidomide and Dexamethasone (DVRd) followed by Autologous Stem Cell Transplant (ASCT) in newly diagnosed multiple myeloma patients.

DETAILED DESCRIPTION:
Multiple myeloma (MM) is a malignant plasma cell disorder characterized by the production of monoclonal immunoglobulin (Ig) proteins or protein fragments (M proteins) that have lost their function.

JNJ-68284528 (ciltacabtagene autoleucel [cilta-cel]) is an autologous chimeric antigen receptor T cell (CAR-T) therapy that targets B-cell maturation antigen (BCMA) that is being evaluated to treat participants with multiple myeloma. The primary hypothesis is that in transplant-eligible participants with newly diagnosed multiple myeloma (NDMM), cilta-cel will significantly improve progression-free survival (PFS) and Sustained MRD-negative CR rate compared with Autologous Stem Cell Transplant (ASCT).

Approximately 750 participants (375 per arm) will be randomly assigned in a 1:1 ratio into 2 arms.

ELIGIBILITY:
Inclusion Criteria:

* Participants with documented NDMM according to IMWG diagnostic criteria, for whom high-dose therapy and ASCT are part of the intended initial treatment plan.
* Measurable disease, as assessed by central laboratory, at screening as defined by any of the following:

  1. Serum monoclonal paraprotein (M-protein) level ≥1.0 g/dL or urine M-protein level ≥200 mg/24 hours; or
  2. Light chain MM without measurable disease in serum or urine: serum Ig free-light chain (FLC) ≥10 mg/dL and abnormal serum Ig kappa lambda FLC ratio.
* ECOG performance status of grade 0 or 1
* Clinical laboratory values within prespecified range.

Exclusion Criteria:

* Prior treatment with CAR-T therapy directed at any target.
* Any prior BCMA target therapy.
* Any prior therapy for MM or smoldering myeloma other than a short course of corticosteroids
* Received a strong cytochrome P450 (CYP)3A4 inducer within 5 half-lives prior to randomization
* Received or plans to receive any live, attenuated vaccine (except for COVID-19 vaccines) within 4 weeks prior to randomization.
* Known active, or prior history of central nervous system (CNS) involvement or clinical signs of meningeal involvement of MM
* Stroke or seizure within 6 months of signing Informed Consent Form (ICF)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 759 (Actual)
Dates: Start 2023-10-10 (Actual); Primary Completion 2033-06 (Estimated); Study Completion 2040-08 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) | up to 10 years ( or 300 PFS events)
  Progression free survival is defined as the time from the date of randomization to the date of first documented PD, as defined in the IMWG criteria, or death due to any cause, whichever occurs first
Sustained MRD-negative CR | up to 24 months
  Sustained MRD-negative CR is defined as being MRD negative by bone marrow aspirate, as determined by NGS with a sensitivity of at least 10-5, and meeting the IMWG criteria for CR, and with MRD-negativity status confirmed at a minimum 12 months apart and without any examination showing MRD-positive status or PD in between.

SECONDARY OUTCOMES:
Overall Response (OR) | up to 17 years
  OR is defined as participants who achieve a partial response (PR) or better according to the IMWG criteria.
Complete Response (CR) or better status | up to 17 years
  CR or better is defined as percentage of participants who achieve a CR response or Stringent Complete Response (sCR) response according to the IMWG criteria.
Overall Minimal Residual Disease (MRD) -negative CR | up to 17 years
  achieving MRD-negative CR, as determined by NGS at any time after the date of randomization before initiation of subsequent antimyeloma therapy.
Time to subsequent antimyeloma therapy | up to 17 years
  Time to subsequent anti-myeloma therapy is defined as the time from randomization to the start of subsequent anti-myeloma therapy.
Progression Free Survival on Next-line Therapy (PFS2) | up to 17 years
  the time from the date of randomization to the date of event, defined as PD as assessed by investigator that starts after the next line of subsequent therapy, or death due to any cause, whichever occurs first.
Overall Survival (OS) | up to 17 years
  Overall survival is measured from the date of randomization to the date of the participant's death.
Change from Baseline in Health-Related Quality of Life (HRQoL) as Assessed by European Organization for Research and Treatment of Cancer Quality-of-life Questionnaire Core 30 (EORTC-QLQ-C30) Scale Score | up to 17 years
  The EORTC QLQ-C30 includes 30 items in 5 functional scales (physical, role, emotional, cognitive, and social), 1 global health status scale, 3 symptom scales (pain, fatigue, nausea/vomiting), and 6 single symptom items (dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial difficulties). The responses are reported using a verbal rating scale. The item and scale scores are transformed to a 0 to 100 scale. A higher score represents greater HRQoL, better functioning, and more (worse) symptoms.
Change from Baseline in Health-Related Quality of Life as Assessed by MySIm-Q Scale Score | up to 17 years
  The MySIm-Q is a disease-specific PRO assessment complementary to the EORTC-QLQ-C30. It includes 17 items with recall period of "7 days" and responses are reported on a 5-point verbal rating scale. Item responses are scored from 0 to 4. Higher scores indicate greater severity/impact.
Change from Baseline in Health-Related Quality of Life as Assessed by European Quality of Life - 5 Dimensions-5 Levels (EQ-5D-5L) Scale Scor | up to 17 years
  The EQ-5D-5L is a generic measure of health status. The EQ-5D-5L is a 5-item questionnaire that assesses 5 domains including mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each of the 5 dimensions is divided into 5 levels of perceived problems, where Level 1: no problem, Level 2: slight problems, Level 3: moderate problems, Level 4: severe problems and Level 5: extreme problems, plus a visual analog scale rating "health today" with anchors ranging from 0 (worst imaginable health state) to 100 (best imaginable health state).
Change from Baseline in Health-Related Quality of Life as Assessed by Patient Global Impression of Symptom Severity (PGIS) Scale Score | up to 17 years
  The PGIS uses 2 items to assess the participant's perception of the severity of their disease symptoms and impact using a 5-point verbal rating scale. Score ranges from 1 (None) to 5 (Very Severe).
Patient-reported Outcomes Version of the Common Terminology Criteria for Adverse Events (PRO-CTCAE) | up to 280 days
  The National Cancer Institute's PRO-CTCAE is an item library of common adverse events experienced by people with cancer that are appropriate for self-reporting. Each symptom selected for inclusion can be rated by up to 3 attributes characterizing the presence/frequency, severity, and/or interference that ranges from 0 to 4 with higher scores indicating higher frequency or greater severity/impact.

CONTACTS AND LOCATIONS:
Locations (105):
- United States (27):
  - University of Arkansas, Little Rock, Arkansas
  - City of Hope, Duarte, California
  - UC San Diego Health Moores Cancer Center, San Diego, California
  - University of California San Francisco (UCSF), San Francisco, California
  - Stanford University, Stanford, California
  - Moffitt Cancer Center, Tampa, Florida
  - Emory University Hospital, Atlanta, Georgia
  - University of Chicago, Chicago, Illinois
  - University of Iowa, Iowa City, Iowa
  - University Of Maryland Medical Center, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Boston Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Karmanos Cancer Center, Detroit, Michigan
  - Mount Sinai Medical Venter, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - University of Rochester, Rochester, New York
  - Montefiore M-E Center, The Bronx, New York
  - Levine Cancer Institute, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - The Ohio State University, Columbus, Ohio
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - University of Virginia, Charlottesville, Virginia
  - Fred Hutchinson Cancer Center, Seattle, Washington
  - Medical College Wisconsin, Milwaukee, Wisconsin
- Australia (9):
  - Princess Alexandra Hospital, Brisbane
  - Royal Prince Alfred Hospital, Camperdown
  - Royal Brisbane and Womens Hospital, Herston
  - Alfred Health, Melbourne
  - Austin Hospital, Melbourne
  - Peter MacCallum Cancer Centre, Melbourne
  - Fiona Stanley Hospital, Murdoch
  - Calvary Mater Newcastle Hospital, Waratah
  - Westmead Hospital, Westmead
- Belgium (4):
  - Jules Bordet Instituut, Anderlecht
  - UZA, Antwerp
  - UZ Gent, Ghent
  - UZ Leuven, Leuven
- Canada (8):
  - Cross Cancer Institute, Edmonton
  - McMaster University, Hamilton
  - Hopital Maisonneuve-Rosemont, Montreal
  - Mcgill University Health Centre, Montreal
  - Ottawa Hospital Research Institute, Ottawa
  - (CHU) Centre Hospitalier Universitaire de Quebec Laval, Québec
  - Princess Margaret Cancer Centre, Toronto
  - Vancouver General Hospital, Vancouver
- Czechia (4):
  - Fakultni nemocnice Brno, Brno
  - Fakultni nemocnice Hradec Kralove, Králová
  - Fakutni nemocnice Ostrava, Ostrava
  - Fakultni nemocnice Plzen, Pilsen
- France (6):
  - CHRU de Lille - Hopital Claude Huriez, Lille
  - Hospices Civils De Lyon, Lyon
  - CHU De Nantes - Hématologie Clinique, Nantes
  - CHU Poitiers - Pôle régional de Cancérologie, Poitiers
  - Hopital Saint Louis - Aphp Hôpitaux Universitaires Saint-Louis, Saint-Louis
  - CHU de Toulouse, Toulouse
- Germany (5):
  - University Hospital of Cologne, Cologne
  - Universitätsklinikum Hamburg - Eppendorf, Hamburg
  - University Hospital of Leipzig, Leipzig
  - Tübingen, Tübingen
  - University Hospital of Würzburg, Würzburg
- Greece (2):
  - Attikon University General Hospital of Attica, Athens
  - 'G. Papanikolaou' Hospital of Thessaloniki, Thessaloniki
- Israel (3):
  - Hadassah Medical Center, Jerusalem
  - Sheba medical center, Ramat Gan
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Japan (10):
  - Kyushu University Hospital - Hematology/Oncology, Fukuoka
  - Hokkaido University Hospital-Department of Hematology, Hokkaido
  - Hyogo College of Medicine, Hyōgo
  - Kanazawa University Hospital, Kanazawa
  - Nagoya City University Hospital - Department of Hematology & Oncology, Nagoya
  - Okayama University Hospital - Hematology/Oncology, Okayama
  - Osaka metropolitan university hospital, Osaka
  - Japanese Red Cross Medical Center - Hematology, Shibuya City
  - Keio University Hospital - Hematology, Shinjuku-Ku
  - Tohoku University Hospital - Hematology, Tōhoku
- Netherlands (5):
  - VU Medisch Centrum, Amsterdam
  - University Medical Center Groningen, Groningen
  - Radboud UMC, Nijmegen
  - Erasmus MC, Rotterdam
  - UMC Utrecht, Utrecht
- Oslo University Hospital Ullevål - Oncology, Oslo, Norway
- Spain (11):
  - Hospital Universitario Ramón y Cajal, Madrid, Madrid
  - Hospital Universitario Germans Trias i Pujol, Badalona
  - Hospital Clinic de Barcelona, Barcelona
  - Instituto Catalán de Oncología, Barcelona
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - CLINICA UNIV. DE NAVARRA, Pamplona, Pamplona
  - Hospital Universitario de Salamanca, Salamanca
  - Hospital de Santiago de Compostela, Santiago de Compostela
  - Hospital Universitario Virgen del Rocío, Seville
  - Hospital Universitario la Fe, Valencia, Valencia
- Sweden (4):
  - Sahlgrenska Universitetssjukhuset, Gothenburg
  - Landstinget i Ostergotland-Universitetssjukhuset i Linkoping, Linköping
  - Skånes University Hospital Lund, Lund
  - Akademiska Sjukhuset, Uppsala
- Switzerland (4):
  - Universitaetsspital Basel - Zentrum fur Hamato-Onkologie, Basel
  - Universitaetsspital Bern, Inselspital, Bern
  - Centre Hospitalier Universitaire Vaudois (CHUV)Département d'oncologie, Lausanne
  - Universitaetsspital Zuerich -Universitaeren Herzzentrum Zuerich, Zurich
- United Kingdom (2):
  - Queen Elizabeth Medical Centre, Birmingham
  - University Hospital of Wales, Cardiff

IPD SHARING:
Plan to Share IPD: No